CLINICAL TRIAL: NCT05913128
Title: Comparison Between Glandular Urethral Disassembly Technique Versus Tubularized Incised Plate Technique for Primary Distal Hypospadius Repair
Brief Title: Comparison Between Glandular Urethral Disassembly Versus Tubularized Incised Plate for Primary Distal Hypospadius Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abou Elezz Abdel Fattah, Lecturer of urology, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rc 7-2-2023
Record Dates: First submitted 2023-03-28; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Glandular Urethral Disassembly; Tubularized Incised Plate; Distal Hypospadius Repair
Keywords: Glandular Urethral Disassembly, Tubularized Incised Plate, Distal Hypospadius

STUDY DESIGN:
Intervention Model Description: Prospective randomized clinical trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First arm (Active Comparator): Glandular Urethral Disassembly technique
  Interventions: Procedure: Glandular Urethral Disassembly technique
- Second arm (Active Comparator): Tubularized Incised Plate technique
  Interventions: Procedure: Glandular Urethral Disassembly technique

INTERVENTIONS:
Procedure: Glandular Urethral Disassembly technique — For Primary Distal Hypospadius Repair
  Other Names: Tubularized Incised Plate technique

SUMMARY:
To compare Glandular Urethral Disassembly technique versus Tubularized Incised Plate technique for Primary Distal Hypospadius Repair

DETAILED DESCRIPTION:
Aim of study to compare glandular Urethral Disassembly technique versus Tubularized Incised Plate technique for Primary Distal Hypospadius Repair

ELIGIBILITY:
Inclusion Criteria:

* Primary Distal Hypospadius

Exclusion Criteria:

* secondary Distal Hypospadius Recurrent Hypospadius

Ages: 6 Months to 6 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 86 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Hospital stay | up to14 days
  Hospital stay will be recorded in days.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed AE Abdel Fattah, PhD, Principal Investigator — faculty of medicine
Locations (1):
- Faculty of medicine, Banhā, Qalyubia Governorate, Egypt